CLINICAL TRIAL: NCT03181945
Title: Comparison of 4 Weeks Versus 12 Weeks Anti-convulsant Therapy for Acute Symptomatic Seizure in Children With Acute Encephalitis Syndrome- Open Label, Randomized Controlled Trial
Brief Title: Duration of Anti-convulsant Therapy for Acute Symptomatic Seizure in Acute Encephalitis Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dhawan Sumeet Rajendra, Senior Resident, Department of Pediatrics, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2016/114
Record Dates: First submitted 2017-06-02; First posted 2017-06-09 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-09

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures | interventions — Population Groups

STUDY DESIGN:
Intervention Model Description: Whether 4 weeks anti-epileptic drug is as efficacious as 12 weeks anti-epileptic drug therapy for Acute Encephalitis syndrome
Masking Description: Open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 4 weeks (Active Comparator): Anti-epileptic drug (as used by treating physician for management of acute symptomatic seizure) for 4 weeks followed by taper in 10-14days
  Interventions: Other: Group 4 weeks
- Group 12 weeks (Active Comparator): Anti-epileptic drug (as used by treating physician for management of acute symptomatic seizure) for 12 weeks followed by taper in 10-14days
  Interventions: Other: Group 12 weeks

INTERVENTIONS:
Other: Group 4 weeks — Anti-epileptic drug (as used by treating physician for management of acute symptomatic seizure) for 4 weeks followed by taper in 10-14days
  Arms: Group 4 weeks
Other: Group 12 weeks — Anti-epileptic drug (as used by treating physician for management of acute symptomatic seizure) for 12 weeks followed by taper in 10-14days
  Arms: Group 12 weeks

SUMMARY:
There are no guidelines or studies evaluating duration of anti-epileptic drugs in central nervous system infections. The duration of anti-epileptic drug is extrapolated from traumatic brain injury in which duration of 1 weeks to 3 months is suggested. So the investigators plan to conduct this study to decide the optimal duration of anti-epileptic drug in acute symptomatic seizure in central nervous system infections

DETAILED DESCRIPTION:
Demography data, seizure details at diagnosis of acute encephalitis syndrome, details of etiology, neuroimaging findings and electroencephalography. A detailed neurological examination will be done in all participants and asked for seizure semiology at admission. Seizure details include seizure type, duration, number of seizures, number of days for which seizures were recurring, status epilepticus, encephalopathy in between seizures. After the initial assessment participants would be randomized into 2 groups: Group 1: Anti-epileptic drug for 4 weeks followed by taper in 10-14days and Group 2: Anti-epileptic drug for 12 weeks followed by tapering over 10-14days. The primary outcome would be be to study the seizure relapse rate (proportion) after stopping anti-epileptic drugs in participants with acute symptomatic seizure given 4weeks and 12 weeks anti-epileptic drug therapy in the two study groups.

Clinical status will be assessed at enrollment as defined by Pediatric Cerebral Performance Category, Pediatric overall Performance Category and Glasgow Outcome Scale-Extended Pediatric Version (GOS-P)

ELIGIBILITY:
Inclusion Criteria:

* Children with acute encephalitis syndrome with acute symptomatic seizures on single anti-epileptic drug will be enrolled in Out patient clinic at 4 weeks of illness

Exclusion Criteria

* Children with chronic meningitis, brain abscess, intracranial Space occupying lesion
* Children with prior history of seizures, prior focal neurological deficit
* Children with abnormal development prior to development of seizures
* HIV, Chronic Liver disease, Chronic Kidney disease, acute hepatic encephalopathy
* Children on two or more than 2 anti-epileptic drugs
* Severely affected children (Pediatric Cerebral Performance Category Scale (PCPC) Score, Pediatric Overall Performance Category Scale with category score of 5)
* Refusal of consent

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-09-30 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Seizure relapse rate | 6 months
  Seizure relapse rate (proportion of participants) developing seizures after randomization

SECONDARY OUTCOMES:
Correlation of EEG findings at time of stoppage of anti-epileptic drug with seizure recurrence | 6 months
  Correlation of EEG at randomization and seizure recurrence will be done
Factors associated with seizure recurrence | 6 months
  Factors associated with seizure recurrence in the two groups
Seizure relapse rate | 12 months
  Seizure relapse rate (proportion of participants) developing seizures after randomization
Seizure relapse rate | 18 months
  Seizure relapse rate (proportion of participants) developing seizures after randomization
Seizure relapse rate | 24 months
  Seizure relapse rate (proportion of participants) developing seizures after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Sumeet Dhawan, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dhawan SR, Sahu JK, Singhi P, Sankhyan N, Jayashree M. Comparison of 4 weeks versus 12 weeks antiseizure medication for acute symptomatic seizures in children with Acute Encephalitis Syndrome: An open-label, randomized controlled trial. Seizure. 2021 Nov;92:182-188. doi: 10.1016/j.seizure.2021.09.005. Epub 2021 Sep 10. PMID 34543779